CLINICAL TRIAL: NCT05770960
Title: Placebo-controlled Crossover Study of the Ability of Naloxegol to Reverse Opioid Effect on Colonic Motor Patterns in Healthy Volunteers
Brief Title: Colonic Motor Patterns in Healthy Volunteers
Acronym: NaloxegolHRM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: S61159
Record Dates: First submitted 2018-08-08; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Opioid-Induced Constipation
Keywords: Naloxegol; Codeine; Colonic manometry; HRM; Motility; Opioid induced constipation; OIC
MeSH Terms: conditions — Opioid-Induced Constipation | interventions — naloxegol; Codeine

STUDY DESIGN:
Intervention Model Description: Randomized double-blind cross-over design (three-way)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Naloxegol - Codeine phosphate (Active Comparator): Participants will receive Naloxegol 25 mg and Codeine syrup in 30 mL and an additional 15 mL at a later stage during the day.
  Interventions: Drug: Naloxegol; Drug: codeine phosphate
- Placebo - Codeine phosphate (Other): Participants will receive Placebo instaid of Naloxegol 25 mg and Codeine syrup in 30 mL and an additional 15 mL at a later stage during the day.
  Interventions: Drug: codeine phosphate; Other: Placebo
- Naloxegol - Placebo (Other): Participants will receive Naloxegol 25 mg and Sirupus simplex syrup (as a placebo alternative for Codeine syrup) in 30 mL and an additional 15 mL at a later stage during the day.
  Interventions: Drug: Naloxegol; Other: Placebo

INTERVENTIONS:
Drug: Naloxegol — Oral administration of Naloxegol after waking up from the Midazolam administration during the colonoscopy.
  Other Names: Movantik; Moventig
  Arms: Naloxegol - Codeine phosphate; Naloxegol - Placebo
Drug: codeine phosphate — Oral administration of Codeine after waking up from the Midazolam administration during the colonoscopy.
  Other Names: Bronchodine
  Arms: Naloxegol - Codeine phosphate; Placebo - Codeine phosphate
Other: Placebo — Oral administration of siripus simplex syrup after waking up from the Midazolam administration during the colonoscopy.
  Other Names: Siripus simplex syrup
  Arms: Naloxegol - Placebo; Placebo - Codeine phosphate

SUMMARY:
Characterization of motor patterns with opioid agonists (codeine) ingestion, and their reversal by a peripherally acting mu-opioid receptor antagonist (Naloxegol).

DETAILED DESCRIPTION:
Opioid induced constipation (OIC) is a highly prevalent condition amongst patients treated with opioids, usually for the treatment of chronic pain, both for malignant and non-malignant causes. The prevalence of constipation and other gastrointestinal side effects among chronic opioid users is 40-90%, depending on the underlying pathology, resulting in non-compliance with pain medication or a reduction in quality of life.

Opioid receptors in the brain are the target for opioids to induce analgesia. Peripheral opioid receptors, mostly μ receptors, are prevalent in the enteric nervous system, and their activation underlies the occurrence of gastrointestinal side effects of opioids. Opioid-agonist binding to enteric μ receptors results in inhibition of gastric emptying, pyloric muscle tone increase, disturbance of the migrating motor complex, delayed bowel transit, decreased intestinal secretions and an elevation of anal sphincter resting pressure.

Peripherally acting μ-opioid receptor antagonists are the treatment of preference for opioid-induced constipation, because they do not cross the blood-brain barrier (BBB) and so do not interfere with central analgesic effects. This peripheral mechanism is the core mechanism of Naloxegol, the most well-known agent for treating opioid overdosing. Through PEGylating, Naloxegol is a P-glycoprotein substrate with very low ability to cross the blood brain barrier (BBB). Studies have shown the ability of Naloxegol improve opioid-induced constipation in patients chronically treated with opioids, not responding to laxatives, significantly. However, the effects of opioids on colonic motor function and their reversal by opioid antagonists are poorly studied.

High-resolution manometry (HRM) of the colon is a sophisticated system for studying colonic motility. Over the last few years, using this approach, it has been possible to differentiate multiple motor patterns. Research is ongoing in different functional bowel disorders (FBDs) to establish the contribution of changes in colonic motor patterns to the disease mechanism and/or symptom generation.

By measuring pressures with HRM during drug administration, we want to gain insight in bowel function and motor pattern changes during treatment. HRM motor pattern analysis will help to substantiate previous findings in bowel function and OIC symptom improvements in OIC patients treated with Naloxegol.(5) We will study colonic motor patterns in healthy volunteers (HV) in a randomized, double-blind, cross-over designed trial with codeine and Naloxegol, using previously established HRM protocols and drug doses.

ELIGIBILITY:
Inclusion Criteria:

1. HV is a man or woman aged 18 to 65 years, inclusive, at prescreening.
2. Normal stool pattern of between 3 defecations per day and 3 per week with a Bristol Stool Form Scale (BSFS) of 1, 2, 6 or 7 in less than 25% of defaecations.
3. HV has not used any opioid medication 14 days prior to randomization.
4. Medications taken for the treatment of allergies, chronic medical conditions, and migraine headaches can be taken during this study (with the exception of opioids for acute treatment of migraines). HV must be on a stable dose of medication for chronic migraines or preventative therapy for at least 1 month at prescreening. HV on stable doses of antidepressants (i.e., for the 3 months prior to prescreening) will be allowed to participate in the study. As needed use of benzodiazepines, if habitual, is permitted.
5. Female subjects must either be:

   1. postmenopausal, defined as 52 years or older and amenorrheic for at least 2 years at prescreening,
   2. surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation, or otherwise be incapable of pregnancy),
   3. abstinent, or
   4. if sexually active, be practicing an effective method of birth control such as hormonal prescription oral contraceptives, progesterone implants or injections, contraceptive patch, intrauterine device, or male partner with a vasectomy.
6. HV must sign an informed consent document before the initiation of any study-related procedures indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study.

Exclusion Criteria:

1. HV has a history of inflammatory or immune-mediated GI disorders including inflammatory bowel disease (ie, Crohn's disease, ulcerative colitis), celiac disease and functional bowel disorder.
2. HV has a history of diverticulitis.
3. HV has a history of intestinal obstruction, stricture, toxic megacolon, GI perforation, gastric banding, bariatric surgery, adhesions, ischemic colitis, or impaired intestinal circulation (eg, aortoiliac disease).
4. HV has any of the following surgical history:

   1. Any abdominal surgery within the 3 months prior to prescreening;
   2. HV has a history of major gastric, hepatic, pancreatic, or intestinal surgery (appendectomy, hemorrhoidectomy, or polypectomy greater than 3 months post-surgery are allowed).
5. HV has current evidence of laxative abuse.
6. HV has a history of a cardiovascular event, including stroke, myocardial infarction, congestive heart failure, or transient ischemic attack within 6 months prior to prescreening.
7. HV has an unstable renal, hepatic, metabolic, or hematologic condition.
8. HV has a history of malignancy within 5 years before prescreening (except squamous and basal cell carcinomas and cervical carcinoma in situ).
9. HV has abnormal thyroid function test as confirmed by thyroid-stimulating hormone <0.3 mcIU/mL or ≥5 mcIU/mL at Prescreening. However, patients who are clinically euthyroid due to thyroid supplement are candidates for the study.
10. HV has current (within 14 days of randomization) or expected use of any narcotic or opioid containing agents, docusate, enemas, GI preparations (including antacids containing aluminum or magnesium, antidiarrheal agents, antinausea agents, antispasmodic agents, bismuth, or prokinetic agents).
11. HV has received an investigational drug or used an investigational medical device within 30 days prior to randomization, or is currently enrolled in an investigational study.
12. HV is pregnant or breastfeeding.
13. HV has any condition that, in the opinion of the investigator, would compromise the well-being of the patient or the study or prevent the HV from meeting or performing study requirements.
14. No smoking on the day of the investigation and the day prior to it.
15. No consumption of grapefruit or grapefruit juice because it can increase Naloxegol plasma levels.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2019-05-09 (Actual); Study Completion 2019-05-09 (Actual)

PRIMARY OUTCOMES:
Overall prevalence of anterograde colonic motor patterns in the different treatment categories. | 3 times for 6 hours
  Observational

SECONDARY OUTCOMES:
Evaluation of the overall prevalence of the other colonic motor patterns (retrograde propagating sequences, simultaneous pressure waves, cyclic propagating sequences, high-amplitude propagating sequences) | 3 times for 6 hours
  Observational
Evaluation of the overall prevalence of high-amplitude propagating sequences after Bisacodyl | 3 times for 6 hours
  Observational and interventional
Evaluation of the colonic motility index in the left, right and sigmoid colon. | 3 times for 6 hours
  Observational
Percentage of Participants reporting Adverse Events (AE). | 3 times for 6 hours
  Observational

CONTACTS AND LOCATIONS:
Overall Officials: Jan Tack, Professor, Principal Investigator — UZ Leuven / KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: Undecided